CLINICAL TRIAL: NCT07383038
Title: The Effect of Mobilization With Movement on Function, Pain, and Joint Position Sense in Patients With Rotator Cuff Lesions: A Double-Blind Randomized Controlled Trial
Brief Title: Effect of Mobilization With Movement in Patients With Rotator Cuff Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Dr, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEU-FTR3
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tears; Physical Disability
Keywords: rotator cuff lesions; Mulligan mobilization; joint position sense
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, parallel-group interventional clinical trial. Eligible participants diagnosed with rotator cuff lesions will be prospectively assigned to one of three intervention arms: Mobilization with Movement (MWM), conventional physiotherapy, or a control group. Allocation to study arms will be performed using a randomization procedure to minimize selection bias and to ensure comparability between groups at baseline.
  Each study group will follow its assigned intervention protocol throughout the intervention period, and participants will remain in the same group for the duration of the study (parallel assignment). Outcomes will be assessed at two time points: before the initiation of the intervention (baseline) and after completion of the intervention period (post-intervention). There will be no crossover between groups.
Who Masked: Investigator
Masking Description: This study will be conducted using a single-blind design. Due to the nature of the manual therapy interventions, it is not feasible to blind participants or treating physiotherapists to group allocation. However, the outcome assessor will be blinded to the participants' group assignments in order to minimize measurement and assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy Group (Active Comparator): Participants in this arm will receive a conventional physiotherapy program commonly used in the conservative management of rotator cuff lesions. The program will include therapeutic exercises, stretching, and physical therapy modalities aimed at reducing pain and improving shoulder function. Mobilization with Movement or other Mulligan-based manual therapy techniques will not be applied in this group.
  Interventions: Other: Conventional Physiotherapy
- Mobilization with Movement (MWM) Group (Experimental): Participants allocated to this arm will receive Mobilization with Movement interventions based on the Mulligan concept. The technique will involve the application of sustained accessory glenohumeral joint mobilization combined with active, pain-free shoulder movements. Interventions will be administered by a trained physiotherapist according to a standardized protocol. This group may also receive basic conventional physiotherapy components excluding other manual mobilization techniques.
  Interventions: Other: Mulligan mobilization
- Control Group (No Intervention): Participants assigned to the control arm will not receive any physiotherapy or manual therapy intervention during the study period. They will undergo the same assessment procedures as the other groups at baseline and post-intervention. After completion of the study, participants in the control group will be offered appropriate rehabilitation if required.

INTERVENTIONS:
Other: Mulligan mobilization — Participants assigned to the Mobilization with Movement (MWM) group will receive manual therapy based on the Mulligan concept. The intervention will consist of the application of sustained, pain-free accessory mobilization to the glenohumeral joint combined with active physiological shoulder movements, primarily in shoulder flexion and abduction. The direction and grade of mobilization will be individually determined according to the patient's symptoms and movement restrictions, ensuring that all movements are performed within a pain-free range.
  MWM interventions will be administered by a trained physiotherapist following a standardized treatment protocol. Each treatment session will last approximately 20-30 minutes and will be applied multiple times per week throughout the intervention period. The primary goal of the intervention is to improve joint mechanics, reduce pain, and enhance proprioceptive input by facilitating normal, pain-free movement patterns.
  Arms: Mobilization with Movement (MWM) Group
Other: Conventional Physiotherapy — Participants allocated to the conventional physiotherapy group will receive a standard rehabilitation program commonly used for rotator cuff lesions. The intervention will include therapeutic exercises targeting shoulder range of motion, strengthening of the rotator cuff and scapular stabilizing muscles, and stretching exercises for periarticular soft tissues. Physical therapy modalities such as heat or ultrasound may be applied as needed for pain management.
  This intervention will be delivered by a physiotherapist according to established clinical guidelines. Mobilization with Movement or other Mulligan-based manual therapy techniques will not be included in this group.
  Arms: Conventional Physiotherapy Group

SUMMARY:
This randomized controlled trial aims to investigate the effects of Mobilization with Movement (MWM) on pain, functional status, and joint position sense in individuals with rotator cuff lesions. Rotator cuff pathology is a common cause of shoulder pain and functional limitation, and impairments in proprioception may further compromise shoulder motor control and recovery.

Eligible participants with rotator cuff lesions will be randomly allocated into three groups: (1) Mobilization with Movement (MWM), (2) conventional physiotherapy, and (3) control group. All participants will be evaluated before and after the intervention period. Outcome measures will include shoulder-related functional disability assessed by the QuickDASH questionnaire, pain intensity, and shoulder joint position sense evaluated using an active repositioning test with a laser pointer during shoulder flexion.

The study is designed to determine whether MWM provides additional benefits over conventional treatment or no intervention in improving pain, function, and proprioceptive accuracy. The findings are expected to contribute to evidence-based conservative rehabilitation strategies for patients with rotator cuff lesions.

DETAILED DESCRIPTION:
Rotator cuff lesions are among the most common causes of shoulder pain and functional limitation, particularly in middle-aged and older adults. Due to the wide range of motion and complex biomechanics of the glenohumeral joint, integrity of the rotator cuff muscles is essential for dynamic stability, coordinated movement, and precise joint positioning. Pathological changes in the rotator cuff may lead not only to pain and reduced functional capacity but also to impairments in proprioception, which can negatively affect motor control and increase the risk of recurrent injury.

Conservative management is widely recommended as the first-line treatment for rotator cuff lesions and typically includes therapeutic exercises, physical agents, and manual therapy techniques. Mobilization with Movement (MWM), developed within the Mulligan concept, is a manual therapy approach that combines sustained accessory joint mobilization with active, pain-free physiological movement. MWM is proposed to improve joint mechanics, reduce pain, and enhance neuromuscular and proprioceptive input. While previous studies have demonstrated the effectiveness of MWM in reducing pain and improving function in various musculoskeletal conditions, evidence regarding its effects on shoulder proprioception, particularly joint position sense, in individuals with rotator cuff lesions remains limited.

This randomized controlled trial is designed to evaluate the effects of MWM on pain, functional outcomes, and joint position sense in patients with rotator cuff lesions. Eligible participants diagnosed with rotator cuff pathology will be randomly assigned to one of three groups: (1) Mobilization with Movement (MWM) group, (2) conventional physiotherapy group, or (3) control group. Randomization will be performed after baseline assessment to ensure allocation concealment.

All participants will undergo standardized assessments at baseline (pre-intervention) and after completion of the intervention period (post-intervention). Functional status of the upper extremity will be evaluated using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire. Pain intensity will be assessed using validated self-report measures. Shoulder proprioception will be assessed through a joint position sense test using an active repositioning method during shoulder flexion with a laser pointer system, recording the deviation from a predefined target point in centimeters.

The MWM group will receive manual therapy interventions based on Mulligan principles, applied by a trained physiotherapist, in addition to standard care. The conventional physiotherapy group will receive commonly used rehabilitation interventions excluding MWM techniques. The control group will not receive therapeutic intervention during the study period. All procedures will be conducted in accordance with the Declaration of Helsinki, and written informed consent will be obtained from all participants prior to enrollment.

The primary objective of this study is to determine whether MWM leads to superior improvements in pain, functional ability, and joint position sense compared with conventional physiotherapy and no intervention. Secondary objectives include evaluating the magnitude of treatment effects and exploring the relationship between changes in proprioception and functional outcomes. The results of this trial are expected to provide clinically relevant evidence regarding the role of Mobilization with Movement in conservative rehabilitation protocols for individuals with rotator cuff lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Clinical and/or imaging-confirmed diagnosis of rotator cuff lesion (e.g., tendinopathy or partial tear)
* Presence of shoulder pain for at least 3 months
* Pain and functional limitation during shoulder movements
* Ability to actively perform shoulder movements required for assessment and intervention
* No physiotherapy or manual therapy treatment for the affected shoulder within the last 3 months

Exclusion Criteria:

* History of shoulder surgery on the affected side
* Full-thickness rotator cuff tear or shoulder instability
* Shoulder fracture, dislocation, or acute trauma within the past 6 months
* Neurological disorders affecting the upper extremity (e.g., cervical radiculopathy, peripheral neuropathy)
* Systemic inflammatory or rheumatologic diseases
* Severe shoulder osteoarthritis or adhesive capsulitis
* Current participation in another clinical trial
* Use of corticosteroid injection in the affected shoulder within the last 3 months
* Pregnancy
* Inability to comply with the study protocol or assessment procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand questionnaire. | Baseline (pre-intervention) and at the end of the 8-week intervention period.
  Upper Extremity Functional Disability, Higher scores better outcomes

SECONDARY OUTCOMES:
Visual Analog Scale | Baseline (pre-intervention) and at the end of the 8-week intervention period.
  Pain Intensity-Lower score better outcomes
Joint Position Sense Error (cm) | Baseline (pre-intervention) and at the end of the 8-week intervention period.
  Shoulder Joint Position Sense-Proprioception was assessed by measuring joint position sense (JPS) using a laser.Lower score better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected in this study will not be made publicly available. Aggregate data and study results will be reported in scientific publications and presentations without including any identifiable participant information.

REFERENCES:
- [Result] Ozlu O, Sahin M. The effect of mulligan mobilization technique application in addition to conventional physiotherapy on pain and joint range of motion in people with neck pain. J Bodyw Mov Ther. 2024 Jul;39:225-230. doi: 10.1016/j.jbmt.2024.02.009. Epub 2024 Mar 5. PMID 38876630